CLINICAL TRIAL: NCT01012232
Title: The Volume-concentration Relationship of Analgesic Efficacy With Intra-capsular Local Anesthetic in Total Knee Arthroplasty: a Randomized, Double-blind, Cross-over Trial.
Brief Title: Local Anesthetic in Total Knee Arthroplasty (TKA): Volume Versus Concentration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundbeck Foundation (Other)
Responsible Party: Lasse Andersen, The Lundbeck Centre for Fast-track Hip and Knee Arthroplasty
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-D-2009-016
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Postoperative Pain; Analgesic Efficacy
Keywords: total knee arthroplasty; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low volume local anesthetic (Active Comparator): bolus injection of local anesthetic in low volume/high concentration (10 mL, 10 mg/mL)
  Interventions: Drug: 10 mL ropivacaine 10 mg/mL
- high volume local anesthetic (Experimental): bolus injection of ropivacaine in high volume/low concentration (20 ml, 5 mg/mL)
  Interventions: Drug: 20 mL ropivacaine 5 mg/mL

INTERVENTIONS:
Drug: 20 mL ropivacaine 5 mg/mL
  Arms: high volume local anesthetic
Drug: 10 mL ropivacaine 10 mg/mL
  Arms: low volume local anesthetic

SUMMARY:
In a randomized, double-blind, cross-over trial, 48 patients scheduled for total knee arthroplasty with placement of an intracapsular catheter will be randomized to receive bolus injection of ropivacaine in high volume/low concentration (20 ml, 5 mg/mL) or low volume/high concentration (10 mL, 10 mg/mL) 6 and 24 hours postoperatively, and pain will be assessed at rest and with mobilization for 2 hours after injections.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for total knee arthroplasty
* Able to give informed oral and written consent to participate

Exclusion Criteria:

* Treatment with opioids or steroids, rheumatoid arthritis or other immunological diseases
* History of stroke or any neurological or psychiatric disease potentially influencing pain perception (e.g. depression, diabetic neuropathy etc.)
* Allergies to any of the drugs administered.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 32 hours postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Lundbeck Centre for fast-track hip and knee arthroplasty, Copenhagen, Denmark